CLINICAL TRIAL: NCT06912100
Title: A Pilot Study of the Probiotic L. Acidophilus (Strain TW01) on Gut Health, Body Composition, and Inflammation
Brief Title: L. Acidophilus (Strain TW01) on Gut Health, Body Composition, and Inflammation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Christopher Blesso, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B2025-0034
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Overweight (BMI > 25); Obese, Otherwise Healthy Volunteers
Keywords: obesity; probiotics; gut health
MeSH Terms: conditions — Overweight; Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo phase (Placebo Comparator): Participants consume capsules containing only an inactive placebo (maltodextrin and magnesium stearate).
  Interventions: Dietary Supplement: Placebo
- Probiotic phase (Experimental): Participants consume capsules containing L. acidophilus (TW01) at 4×10^10 CFU/capsule (three capsules daily, totaling 1.2×10^11 CFU/day) plus a commercial fiber source (Fibersol-2).
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Placebo — Participants consume capsules containing only an inactive placebo (maltodextrin and magnesium stearate).
  Arms: Placebo phase
Dietary Supplement: Probiotic — Participants consume capsules containing L. acidophilus (TW01) at 4×10^10 CFU/capsule (three capsules daily, totaling 1.2×10^11 CFU/day) plus a commercial fiber source (Fibersol-2).
  Arms: Probiotic phase

SUMMARY:
This is a pilot research study to investigate the effects of a probiotic supplement (L. acidophilus, strain TW01) on substances found in the stool and bloodstream, gut bacteria composition, body composition, as well as any relationship of these substances with markers of inflammation. Lactobacillus acidophilus is commonly found in a variety of fermented foods, including yogurt, cheese, and kefir, due to its ability to produce lactic acid and other substances. This bacterium is generally well-tolerated in healthy individuals and has a longstanding history of safe use. The investigators are doing this pilot study to see if a particular probiotic, called L. acidophilus (strain TW01) and isolated from fermented coffee grounds, can make a positive difference in human gut and overall health. Specifically, the investigators want to look at how this probiotic affects certain substances in human stool and blood, the makeup of the bacteria in the gut, and aspects of body composition. The investigators are also interested in whether these changes relate to markers of inflammation, which can tell us more about their impact on overall health. This probiotic strain has been shown in other studies to be safe and well tolerated, and the investigators hope our research will help us better understand how it works and whether it might support health in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years
2. Body mass index (BMI) between 28 kg/m2 and 40 kg/m2
3. Waist circumference ≥ 88 cm or 35 inches for women, ≥ 102 cm or 40 inches for men
4. Willing to consume experimental capsules daily
5. Willing to prepare and consume the delivered meal kits
6. Do not fit any exclusion criteria

Exclusion Criteria:

1. Self-reported history of immunodeficiency, major gastrointestinal surgery, renal or liver disease, diabetes, heart disease, stroke, peripheral artery/vascular disease, cancer, eating disorders, gut-associated pathologies, autoimmune diseases, pacemaker, thyroid disease, gallbladder disease, chronic inflammatory diseases, scleroderma, blood clotting disorders, intravenous drug use
2. Weight changes > 10% over the last 4 weeks
3. Oral antibiotics and/or probiotics use up to 1 month prior to study and during study
4. Currently taking GLP-1 analogues (e.g., Ozempic), anti-inflammatory medications (e.g., corticosteroids), daily use of nonsteroidal anti-inflammatory drugs (NSAIDs) (occasional use is permitted), medications which primarily affect blood clotting (e.g., warfarin), or any medications that suppress the immune system.
5. Dairy allergy
6. Currently pregnant or breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Fecal butyrate | From baseline to the end of each 6-week intervention phase
  Determine the effects of the probiotic on the short-chain fatty acid, butyrate (mmol/L), a marker of gut health in stool

SECONDARY OUTCOMES:
Serum inflammation marker | From baseline to the end of each 6-week intervention phase
  Determine the effects of the probiotic on a marker of inflammation, high-sensitivity C-reactive protein (hsCRP) (mg/L), in the bloodstream
Body fat composition | From baseline to end of each 6-week intervention phase
  Determine the effects of the probiotic on body fat composition by bioelectric impedance analysis (% of body weight).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Department of Nutritional Sciences, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP